CLINICAL TRIAL: NCT00953537
Title: Multicentric Pilot Study of Dihydropyrimidine Dehydrogenase (DPD) Deficiency for Predicting Capecitabine Toxicity in Breast Cancer Patients
Brief Title: Predicting Response to Capecitabine in Women With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000638377; CALACASS-DPD-Sein; 2008/21; INCA-RECF0942; EUDRACT-2008-004136-20
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

ARMS (1):
- capecitabine (Other)
  Interventions: Drug: capecitabine; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: capecitabine
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Identifying genes that increase a person's susceptibility to side effects caused by capecitabine may help doctors plan better treatment.

PURPOSE: This clinical trial is studying blood samples in predicting response to capecitabine in women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the sensitivity, specificity, and positive and negative predictive values of dihydrouracil/uracil (UH_2/U) ratio measured before starting treatment on grade 3-4 capecitabine-related toxicity in women with metastatic breast cancer.

Secondary

* To prospectively test the value of the germinal genotype of thymidylate synthase (TS) and methylenetetrahydrofolate reductase (MTHFR) as predictors of resistance to capecitabine.
* To evaluate the practical feasibility of such pre-therapeutic screening.
* To determine the sensitivity, specificity, and positive and negative predictive values of dihydropyrimidine dehydrogenase genotyping on grade 3-4 capecitabine-related toxicity in the first and second courses.
* To evaluate the predictive gain provided by genotyping relative to phenotyping alone.
* To evaluate the influence of TS and MTHFR gene polymorphisms on clinical response and duration of response.
* To evaluate the pharmacokinetics of capecitabine and its metabolites and their relationship with UH_2/U and genotype.
* To evaluate the total cost of pre-therapeutic phenotyping alone and the combination of phenotyping and genotyping.
* To exhaustively analyze the 23 exons of the dihydropyrimidine dehydrogenase (DPYD) gene in patients who developed toxicity.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected 8-15 days before the start of treatment and periodically on the first day of treatment for dihydropyrimidine dehydrogenase phenotyping (dihydrouracil/uracil ratio and high performance liquid chromatography analysis), genotyping (4 most relevant single nucleotide polymorphisms), and pharmacokinetic analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiologically (by scintography) or histologically confirmed metastatic breast cancer
* At least 1 measurable or evaluable target lesion
* Receiving capecitabine as monotherapy or with targeted antiangiogenic therapies (e.g., bevacizumab or trastuzumab)
* No uncontrolled brain metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Life expectancy ≥ 3 months
* Fertile patients must use effective contraception
* No chronic uncontrolled illness
* No congestive heart failure
* No peripheral venous disease
* No severe uncontrolled infection
* No hypoxemic respiratory failure
* No prior primary cancer except for basal cell carcinoma of the skin
* No psychologic disorder

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No capecitabine co-administered with chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Capecitabine-related toxicity (i.e., hematological, diarrhea, and hand-foot syndrome) recorded during the first and second courses | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Ferrero, MD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France